CLINICAL TRIAL: NCT05473351
Title: Thirst in the Intensive Care Unit, Recognition, Sensitivity and Type
Acronym: THIRST
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220789
Record Dates: First submitted 2022-07-12; First posted 2022-07-25 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Thirst in Intensive Care Unit (ICU) Practice
Keywords: Thirst; Intensive care unit,; Cohort
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thirst: Patients undergoing invasive mechanical ventilation for at least 24 hours in one of the participating centers
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Visual Analogic Scale

SUMMARY:
Thirst is a perception that provokes the desire to drink liquids. It is a multidimensional symptom that is described in terms of intensity and distress and is associated with dry mouth, called xerostomia.

Thirst is poorly recognized in intensive care unit practice. Yet, research has shown that it is one of the most prevalent, most intense, and least well treated symptoms in intensive care patients. Thirst and dry mouth are associated with physical discomfort in the ICU. However, thirst often goes unnoticed and untreated.

In this context, The investigators aim to conduct a prospective observational study in mechanically ventilated patients able to communicate to better understand the prevalence, intensity, mechanisms and prognostic value of thirst as well as dry mouth sensation.

Primary objective: to assess thirst in mechanically ventilated patients. Primary endpoint: visual analog thirst scale from 0 mm (no thirst) to 100 mm (maximal thirst)

1. Patient 18 years of age and older
2. Patients undergoing invasive mechanical ventilation for at least 24 hours at one of the participating centers
3. No objection to participation in the study During the study period, patients from 3 resuscitation sites are systematically screened for inclusion in the study on a daily basis, between 9:00 am and 12:00 pm.

Subjects meeting the inclusion and non-inclusion criteria (with the exception of the delirium test) will be informed of the study by the principal investigator or any other investigator trained and declared in the research. The oral information will be completed by the delivery of an information note. Patients who wish to participate in the study will be given up to 24 hours to consider their decision.

If the patient agrees to participate in the study, his or her non-opposition is collected by the investigator on a dedicated form in duplicate. One copy will be given to the patient, and the other will be kept in the department with the research documents.

In case of suspected confusion, a delirium screening test (CAM-ICU) will be performed to verify the patient's eligibility. If the test confirms the presence of confusion, the patient will be excluded from the study.

The information and the collection of the non-opposition will be notified in the patient's medical file.

Following their inclusion, patients are assessed only once during their stay in the ICU: the day of inclusion.

Once enrolled, patients are asked to rate the intensity of thirst by placing a cursor on a 100 mm visual analog scale (VAS) bounded on the left by "not thirsty" and on the right by "intolerably thirsty".

If a patient understands the principle of the assessment but is unable to move the VAS cursor himself, the observer assists the patient by holding the scale and supporting the patient's forearm. If the subject is unable to move his or her arms (as in some cases of severe neuromuscular impairment), observers are allowed to manipulate the VAS slider following the patient's instructions. However, this is not recommended and should be avoided whenever possible. The slider should never be adjusted directly or solely by the investigator.

The visual analog scales for dry mouth, anxiety, pain and dyspnea will be performed as part of the protocol after the thirst assessment.

The oral status, the search for edema or skin folds and the Revised Oral Assessment Guide (ROAG) score for intubated patients will also be performed at the same time.

An average of 20 minutes is necessary to perform all these procedures.

DETAILED DESCRIPTION:
Thirst was reported in 70% of symptom assessments of intensive care patients. Thirst is a major source of physical discomfort. This should make it a concern for clinicians and ICU nurses whose mission is to alleviate symptoms in addition to treating pathology.

Balancing extracellular and intracellular volume is a goal in the poorly communicating patient with no spontaneous access to water. Thirst may exist, persist, reappear, or increase again after the institution of water intake; it may reveal changes in the intra/extra sector or inappropriate intakes. Thirst could therefore be useful as a clinical management tool. However, it has not been studied to any great extent in mechanically ventilated patients.

Neglecting thirst in these circumstances is bound to cause suffering. This neglect may also offset the physiological benefits in terms of clinical outcomes. It could also have a negative impact at a distance through negative memories. Nevertheless, thirst is not routinely assessed in ICU patients, except after extubation when the patient has access to spontaneous hydration.

Mechanically ventilated patients have multiple causes of thirst and dry mouth and at the same time have difficulty communicating and limited access to water. It is essential to study thirst in this population. In particular, determining the prevalence of thirst in this population would raise awareness of its screening. Finally, understanding the main mechanisms involved in thirst in patients undergoing invasive mechanical ventilation would allow the development of therapeutic solutions to minimize it.

In this context, the investigators wish to conduct a prospective observational study in mechanically ventilated patients able to communicate in order to better understand the prevalence, intensity, mechanisms and prognostic value of thirst as well as the sensation of dry mouth. They will also focus on the relationship of thirst with dyspnea, anxiety and pain.

Description of the study population and rationale for its selection The management of thirst is usually ensured by free access to water and balancing the patient's extracellular volume.

In the mechanically ventilated patient, this management is made more difficult by many factors: lack of free access to water, difficulty in communication, sensation of dry mouth induced by the mechanical ventilation device.

The population studied corresponds to patients under invasive mechanical ventilation in three intensive care units of university hospitals:

Pitié Salpêtrière intensive care medicine unit, Avicenne hospital intensive care medicine unit, and Saint-Louis hospital intensive care medicine unit.

Justification of the duration of the research The objective would be to include 200 patients at a rate of approximately 66 patients per service.

Eligibility criteria Recruitment will consist in considering any patient under mechanical ventilation and communicating as potentially eligible, provided that they meet the inclusion/non-inclusion criteria.

Conduct of the research During the study period, patients from the 3 resuscitation sites are systematically screened for inclusion in the study on a daily basis, between 9:00 am and 12:00 pm.

Subjects meeting the inclusion and non-inclusion criteria will be informed of the study by the principal investigator or any other investigator trained and declared in the research. The oral information will be supplemented by an information note. Patients who wish to participate in the study will be given up to 24 hours to consider their decision.

If the patient agrees to participate in the study, his or her non-opposition is collected by the investigator on a dedicated form in duplicate. One copy will be given to the patient, and the other will be kept in the department with the research documents.

In case of suspected confusion, a delirium screening test (CAM-ICU) will be performed to verify the patient's eligibility. If the test confirms the presence of confusion, the patient will be excluded from the study.

The information and the collection of the non-opposition will be notified in the patient's medical file.

Once recruited, patients are asked to rate the intensity of thirst by placing a cursor on a 100 mm visual analog scale (VAS) bounded on the left by "not thirsty" and on the right by "intolerably thirsty".

If a patient understands the principle of the assessment but is unable to move the VAS cursor himself, the observer assists the patient by holding the scale and supporting the patient's forearm. If the subject is unable to move his or her arms (as in some cases of severe neuromuscular impairment), the observers are allowed to manipulate the VAS slider by following the patient's instructions. However, this is not recommended and should be avoided whenever possible. The slider should never be adjusted directly or solely by the investigator.

Visual analog scales for dry mouth, anxiety, pain, and dyspnea will be performed as part of the protocol after the thirst assessment. The oral status, the search for edema or skin folds and the Revised Oral Assessment Guide (ROAG) score for intubated patients will also be performed at the same time.

Follow-up of the population The included patients are evaluated only once during their stay in the ICU: the day of inclusion. The duration of their participation is estimated at 20 minutes.

Conduct in the presence of thirst in the patient In the event that the patient is thirsty, the investigator will immediately inform the patient's physician.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 18 years of age and older
2. Patients undergoing invasive mechanical ventilation for at least 24 hours at one of the participating centers
3. No objection to participation in the study

Exclusion Criteria:

Exclusion Criteria :

1. Patients unable to communicate verbally and reliably self-report thirst:

   * Richmond Agitation-Sedation Scale (RASS) < -2 or > +2,
   * delirium according to the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) (if confusion is suspected)
   * severe cognitive impairment or severe mental illness
   * non-French speaking patients
   * severe hearing loss.
2. Pregnant women
3. Adults under legal protection
4. Not affiliated to a social security system or not benefiting from such a system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on invasive mechanical ventilation, admitted to one of the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
:Assessment of thirst in mechanically ventilated patients. | Through study completion, an average of 1 year
  visual analog thirst scale from 0 mm (no thirst) to 100 mm (maximum thirst)

SECONDARY OUTCOMES:
Evaluation of the association between thirst and dry mouth in mechanically ventilated patients. | Through study completion, an average of 1 year
  Visual analog scale of dry mouth
Evaluation of the association between thirst and oral status in mechanically ventilated patients. | Through study completion, an average of 1 year
  Oral status: Oral Health Assessment Tool
valuation of the association between thirst and extracellular volume in ventilated patients | Through study completion, an average of 1 year
  Physical examination oriented towards the evaluation of extracellular and intracellular volume: presence of edema of the lower limbs or lumbar region, presence of a skin fold
Evaluation of the association between thirst and anxiety in the mechanically ventilated patient. | Through study completion, an average of 1 year
  Visual Anxiety Scale
Evaluation of the association between thirst and pain in mechanically ventilated patients. | Through study completion, an average of 1 year
  Visual Analogue Pain Scale measures pain intensity. It consists of a 10 numerical values, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Evaluation of the association between thirst and dyspnea in mechanically ventilated patients.ventilated patients. | Through study completion, an average of 1 year
  Visual analog scale of dyspnea measures dyspnea severity. It consists of a 10 numerical values, with two end points representing 0 ('absence of dyspnea') and 10 ('maximum dyspnea')

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service de médecine intensive et réanimation, hôpital Avicenne, Bobigny
  - Service de médecine intensive et réanimation, hôpital Saint-Louis, Paris
  - Service de medecine intensive et réanimation, hôpital Pitié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal